CLINICAL TRIAL: NCT00206440
Title: Evaluation of the Efficacy of Esomeprazole in Suppressing Nausea and Vomiting in Patients Undergoing Chemotherapy for Breast Cancer
Brief Title: Nexium Study To Suppress Nausea During Chemotherapy
Acronym: NEXIUM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Accrual was not optimized
Sponsor: Baylor Breast Care Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Mothaffar Rimawi, Medical Director, Baylor Breast Care Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-16348; Nexium Study (Other: Baylor College of Medicine)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-03-07 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Nausea
Keywords: chemotherapy; nausea; vomiting; breast cancer
MeSH Terms: conditions — Nausea; Vomiting; Breast Neoplasms | interventions — Esomeprazole; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esomeprazole (Experimental): Patients receiving chemotherapy (anthracycline-based) will be randomized to esomeprazole for Cycle 1 Days 1-5 and Cycle 2 Days 1-5
  Interventions: Drug: esomeprazole
- Sugar pill (Placebo Comparator): Subjects will be given placebo Cycle 1 Days 1-5 and Cycle 2 Days 1-5.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: esomeprazole — nexium
  Other Names: nexium
  Arms: Esomeprazole
Other: Placebo — Placebo 1 pill daily Cycle 1 Days 1-5 and Cycle 2 Days 1-5
  Other Names: Sugar Pill
  Arms: Sugar pill

SUMMARY:
This study will look at a drug called esomeprazole, the newest PPI, as a way to further reduce the amount of nausea and vomiting seen in breast cancer patients receiving adriamycin or epirubicin chemotherapy. Esomeprazole may help protect the gut lining from the stomach acid and thus lessen the nausea and vomiting. If patients have less stomach sickness, they may be able to enjoy their daily routines much more while they are getting chemotherapy.

DETAILED DESCRIPTION:
1. Breast Cancer

   The American Cancer Society estimates that there will be approximately 215,990 new cases of breast cancer diagnosed in women during 2004 in the United States. Breast cancer is the most common malignancy in women in the United States and the second leading cause of cancer death in women.

   Treatment options for breast cancer have evolved from extensive surgical approaches to breast-conserving techniques and the use of adjuvant and neo-adjuvant chemotherapy, radiation, and endocrine therapy to reduce the risk of recurrence.
2. Chemotherapy in Breast Cancer

   The use of adjuvant chemotherapy is a well established and routine part of care for breast cancer. Chemotherapy can reduce a woman's risk of recurrence by 25-30%. The amount of risk reduction depends on the patient's age, nodal status, and hormone receptor status.

   Anthracycline-based chemotherapy is standard in the treatment of breast cancer with doxorubicin being the most frequently used agent in this group. Currently the most commonly used chemotherapy regimens for breast cancer include: * doxorubicin/cyclophosphamide (AC) * fluorouracil/doxorubicin/cyclophosphamide (FAC) * cyclophosphamide/methotrexate/fluorouracil (CMF) * docetaxel/doxorubicin/cyclophosphamide (TAC) * fluorouracil/epirubicin/cyclophosphamide (FEC) * single agent taxanes (paclitaxel and docetaxel) Except for the taxanes, these agents are known to cause significant nausea and vomiting after administration.

   Cancer drugs differ both quantitatively and qualitatively in their emetogenic potential. Emetogenic potential can be influenced by chemotherapy-related characteristics and patient characteristics.
3. Gastrointestinal Side Effects of Chemotherapy

Nausea and vomiting following administration of chemotherapy for cancer are among the most significant and feared side effects of patients undergoing treatment. Despite continued advances in pharmacology, the ability to prevent or control nausea, vomiting, or retching remains a problem for patients. Research has confirmed that chemotherapy related nausea and vomiting negatively affects quality of life. Among patients, the same level of nausea and vomiting varies in effect on quality of life. It is difficult to substantiate the degree of this effect, but it has been shown that even with serotonin antagonists, patients still rank nausea as their most bothersome chemotherapy side effect, while vomiting is ranked as third to fifth most bothersome.

The risk for chemotherapy induced nausea and vomiting is related to the anti-neoplastic agents administered and to patient related factors. Emetogenic potential is affected by the intrinsic emetogenicity of the chemotherapy drugs, the combination of agents, the doses administered and the rate of administration. Patient related factors include: 1. gender-increased risk in females 2. age-increased risk in younger, premenopausal patients 3. history of alcohol intake-low chronic intake decreases risk 4. history of motion sickness-increases risk 5. hyperemesis during pregnancy-increases risk.

Emesis is a complex phenomenon characterized by three components: nausea, vomiting, and retching. Nausea is a subjective phenomenon of an unpleasant sensation in the epigastrium and in the back of the throat that may or may not culminate in vomiting; it is also described as feeling "sick at the stomach." Nausea exists only insofar as it is defined by the patient. Vomiting is the forceful expulsion of the contents of the stomach, duodenum and jejunum through the oral cavity as a result of changes in intrathoracic positive pressure. It is also described as "throwing up." Retching, also called "dry heaves," is the attempt to vomit without expelling any material.

Drugs used to improve the control of nausea and vomiting include serotonin antagonists, dopamine antagonist (metoclopramide, prochlorperazine), corticosteroids, benzodiazepines, and phenothiazines. The American Society of Clinical Oncology (ASCO) has developed clinical practice guidelines for the management of chemotherapy-induced nausea and vomiting based on the emetogenic potential of the agents being administered. For combinations with moderate emetogenic potential, acute emesis is managed with a corticosteroid and serotonin receptor antagonists. Serotonin receptor antagonists currently available include ondansetron, granisetron, and dolasetron. Studies indicate they are equally effective in the management of chemotherapy-related nausea/vomiting/retching. Delayed emesis (greater than 24 hours post-chemotherapy) can be controlled with a number of agents including steroids, serotonin receptor antagonists or metoclopramide. Recommended combinations include dexamethasone, 8 mg for 2-3 days, then 4 mg for 1-2 days and metoclopramide, 20-40 mg twice daily to four times daily for 3-4 days, or Zofran 8 mg twice daily for 3 days. With combination chemotherapy, patients should receive the antiemetic regimens appropriate for the chemotherapy agent with the highest emetic risk.

Drugs used to improve the control of nausea and vomiting include serotonin antagonists, dopamine antagonist (metoclopramide, prochlorperazine), corticosteroids, benzodiazepines, and phenothiazines. The American Society of Clinical Oncology (ASCO) has developed clinical practice guidelines for the management of chemotherapy-induced nausea and vomiting based on the emetogenic potential of the agents being administered. For combinations with moderate emetogenic potential, acute emesis is managed with a corticosteroid and serotonin receptor antagonists. Serotonin receptor antagonists currently available include ondansetron, granisetron, and dolasetron. Studies indicate they are equally effective in the management of chemotherapy-related nausea/vomiting/retching. Delayed emesis (greater than 24 hours post-chemotherapy) can be controlled with a number of agents including steroids, serotonin receptor antagonists or metoclopramide. Recommended combinations include dexamethasone, 8 mg for 2-3 days, then 4 mg for 1-2 days and metoclopramide, 20-40 mg twice daily to four times daily for 3-4 days, or Zofran 8 mg twice daily for 3 days. With combination chemotherapy, patients should receive the antiemetic regimens appropriate for the chemotherapy agent with the highest emetic risk.

Studies done with standard antiemetics in women undergoing treatment with anthracycline-based chemotherapy for breast cancer show a success rate for emetic control in the range of 60-65%. 4. Measurement of Nausea, Vomiting, and Retching

It remains difficult to compare clinical studies of nausea and vomiting because of the variety of measurement tools utilized and the variable time periods that were monitored following chemotherapy. The ideal tool would include assessment of: 1. duration and severity of nausea 2. frequency, duration, and severity of vomiting/retching 3. number of antiemetics utilized 4. impact of nausea and vomiting on quality of life 5. adverse effects experienced

5. Proton Pump Inhibitors

Despite utilization of the antiemetics recommended by ASCO, approximately one-third of patients undergoing anthracycline-based chemotherapy still develop nausea and vomiting. A current therapeutic challenge is to find and prove methods to control nausea and vomiting after chemotherapy.

Although the pathophysiology of nausea and vomiting is not well understood, we know that chemotherapy causes damage to the gastrointestinal (GI) mucosa. The pathobiology of the mucosal damage has been reviewed by Blijlevens and can be divided into four phases: the inflammatory phase, the epithelial phase, the ulcerative/bacteriological phase and the healing phase. This mucosal injury is usually self-limiting with a complete cycle of injury to healing lasting approximately 2-3 weeks. The mucosal damage can be increased in patients receiving chemotherapy and corticosteroids which breast cancer patients require as pre-medications. Since cytotoxic chemotherapy damages the mucosal lining, it leaves the GI mucosa exposed to the normal acid-producing gastric parietal cells. The resultant damage has been seen endoscopically in patients receiving chemotherapy with cytosine arabinoside. Hence, suppression of acid secretion from the gastric parietal cells should reduce mucosal injury and related symptoms.

Historical therapies for gastrointestinal distress have included anticholinergics, as well as H-2 receptor antagonists, to help reduce acid secretion. H-2 receptor blockers were effective by blocking the histamine driven acid secretion, but despite its targeted action, acid production continues through alternative pathways. Recently a group of new agents known as proton pump inhibitors have been developed which target the final common pathway of acid secretion. These agents are known to act directly on the H+/K+-ATPase in the gastric parietal cell. Since these agents act directly on the final stimulatory pathway, they provide rapid symptom resolution and reliable healing in gastroesophageal reflux disease and peptic ulcer disease.

To date, two large clinical trials have been performed to evaluate the effectiveness of proton pump inhibitors in preventing mucosal injury. The first trial selected 182 patients with breast cancer (77 pts) or colon cancer (105 pts) who were receiving cyclophosphamide, methotrexate and 5-FU (CMF), or 5-FU, respectively. These patients were randomized to receive either omeprazole (20 mg daily), misoprostol (a prostaglandin analogue) (400 mg twice daily), or placebo (once daily) for two full courses of chemotherapy (56 days). Endoscopic evaluation (EGD) was performed one week prior to initiation of chemotherapy and one week after the end of the second cycle of chemotherapy comparing the number of erosions/ulcers in the stomach and duodenum. The omeprazole group had a lower frequency and degree of erosions compared to placebo and misoprostol. Symptoms of epigastric pain and heartburn were also significantly less in the omeprazole patients. A second study performed by the same group evaluated patients with breast or colon cancer (n=228) receiving either CMF or 5-FU. These patients were randomized to receive omeprazole 20 mg daily, ranitidine 300 mg daily (a H2 blocker), or placebo once daily for 56 days. EGD was performed as above, before cycle 1 and after cycle 2 of chemotherapy. The omeprazole group experienced the lowest frequency of ulcers (n=2), followed by the ranitidine group (n=8), and the placebo group (n=18). Symptoms of epigastric pain or heartburn were also significantly less in the omeprazole arm (n=11) compared to the ranitidine (n=13) or placebo (n=24) arms. Chemotherapy was delayed in the placebo and ranitidine group, but not in the patients receiving omeprazole. These two trials demonstrate the ability of a proton pump inhibitor (omeprazole) to limit the mucosal injury induced by chemotherapy. Protecting the mucosa from damage also appeared to significantly decrease the frequency of upper GI symptoms. It should be noted that nausea or vomiting was not assessed in either trial since various antiemetics were given during chemotherapy.

Esomeprazole magnesium is the latest proton pump inhibitor that has been developed. It is unique in that it is the S- isomer of omeprazole, and as such, has better bioavailability and elevated levels compared to the racemic omeprazole. Since the proton pump is the last step in acid production, blockade of this pump causes reduction in gastric acidity. This effect is dose related up to a dose of 20-40mg daily. Esomeprazole is currently clinically indicated for the treatment of erosive esophagitis and symptomatic gastroesophageal reflux disease. In addition, it is approved to treat Helicobacter pylori in patients with duodenal ulcer disease in conjunction with either amoxicillin or clarithromycin and amoxicillin.

ELIGIBILITY:
Inclusion Criteria:

For inclusion, participants must:

* be female, age 18 years or older
* sign an informed consent
* have Stage I, II, or III breast cancer
* be receiving at least four cycles of anthracycline-based chemotherapy which may include: doxorubicin/cyclophosphamide AC),5-fluorouracil/doxorubicin/cyclophosphamide (FAC), fluoruracil/epirubicin/cyclophosphamide (FEC) or dose dense chemotherapy regimen (AC every two weeks) as their agents for neoadjuvant or adjuvant chemotherapy
* patient must receive a serotonin receptor antagonist and a steroid for premedication
* have a negative serum pregnancy test within 7 days prior to starting study if pre-menopausal
* have adequate renal function, defined by a serum creatinine within 1.5 times the upper limit of normal
* have adequate liver function, defined by a total bilirubin, SGOT, alkaline phosphatase and albumin within 1.5 times the upper limits of normal
* have adequate bone marrow function, defined as a WBC >4.0, platelet count >100K, and HCT >30
* have no prior or current malignancies for which chemotherapy was utilized
* have a performance status of at least 2 according to the Eastern Cooperative Oncology Group World Health Organization or a Karnofsky score of 50% or greater.

Exclusion Criteria:

* pregnancy or unwillingness to use a reliable contraceptive method in women of child-bearing potential
* severe or underlying chronic illness or disease
* renal insufficiency or liver abnormalities
* chronic use of steroids
* uncontrolled GERD
* current use of proton pump inhibitors
* history of Barrett's esophagus
* history of erosive gastritis
* intolerance to serotonin receptor antagonists
* current use of aprepitant or palonosetron as antiemetics
* concomitant use of H2-receptor antagonists (ranitidine, cimetidine, famotidine or nizatidine) or metaclopramide

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-08; Primary Completion 2009-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor Breast Center
Locations (1):
- Baylor Breast Center, Houston, Texas, United States

REFERENCES:
- See also: Web site — http://www.breastcenter.tmc.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Esomeprazole: Subjects will be given esomeprazole 40mg daily by mouth for Cycle 1 Days 1-5 and Cycle 2 Days 1-5.
- Sugar Pill: Subjects will be given placebo(surgar pill) 40mg daily by mouth for Cycle 1 Days 1-5 and Cycle 2 Days 1-5.
Period: Overall Study
Arm/Group | Esomeprazole | Sugar Pill
Started | 21 | 22
Completed | 16 | 18
Not Completed | 5 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Adverse Event | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Sugar Pill | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Customized [Number; unit: participants]
  <40 years | 2 | 3 | 5
  Between 40 and 49 years | 4 | 6 | 10
  Between 50 and 59 years | 11 | 8 | 19
  Between 60 and 69 years | 4 | 3 | 7
  >=70 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Times a Subject Felt Sick to Her Stomach and Number of Times a Subject Required Rescue Medication
Description: Proportion of patients who exhibit no more than one emetic episode and who do not require rescue medication for nausea from 2-7 days following chemotherapy. Thus, we will look at esomeprazole when used to decrease the incidence,severity and duration of nausea/vomiting/retching in breast cancer patients who are receiving anthracycline-based chemotherapy.
Time Frame: 2-7 days following chemotheraphy
Measure: Number; unit: Proportion of patients who exhibit no mo
Groups:
- Esomeprazole: The first dose of esomeprazole 40 mg will be administrated prior to the initiation of chemotherapy along with the standard antiemetics for each cycle. On day 2 to 5 following chemotherapy, the patient will take one capsule each morning.
- Sugar Pill: The frist dose of sugar pill 40 mg will be administrated prior to the initiation of chemotherapy along with the standard antiemetics for each cycle. On day 2 to 5 following chemotherapy, the patient will take one capsule each morning.
Arm/Group | Esomeprazole | Sugar Pill
Number analyzed (Participants) | 20 | 20
Proportion of patients who exhibit no mo
  cycle 1 | 0.8 | 0.8
  cycle 2 | 0.94 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the subjects was enrolled to the study, during the study treatment, and followed up 30 days after termination from the study.
Groups:
- Esomeprazole: The frist dose of esomeprazole 40 mg will be administrated prior to the initiation of chemotherapy along with the standard antiemetics for each cycle. On day 2 to 5 following chemotherapy, the patient will take one capsule each morning.
Arm/Group | Esomeprazole | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 15/21 | 16/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esomeprazole (N=21) | Sugar Pill (N=22)
belching (Gastrointestinal disorders) | 3 (3) | 0 (0)
bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
decreased appetite (Gastrointestinal disorders) | 1 (2) | 0 (0)
fatigue (General disorders) | 4 (4) | 3 (3)
gas (Gastrointestinal disorders) | 2 (2) | 0 (0)
headache (General disorders) | 7 (11) | 8 (10)
mild nausea (Gastrointestinal disorders) | 4 (4) | 3 (4)
nausea (Gastrointestinal disorders) | 4 (6) | 7 (10)
severe nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
taste changes (Gastrointestinal disorders) | 1 (2) | 0 (0)
tiredness (General disorders) | 1 (2) | 0 (0)
vomiting (Gastrointestinal disorders) | 3 (3) | 2 (3)
constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (4)
heartburn (Gastrointestinal disorders) | 0 (0) | 2 (2)
mild fatigue (General disorders) | 0 (0) | 2 (2)
mild headache (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes